CLINICAL TRIAL: NCT01501903
Title: Randomized Trial Comparing the Standard and Fanning Techniques for Fine Needle Aspiration of Pancreatic Mass Lesions at Endoscopic Ultrasound
Brief Title: Standard Versus Fanning Techniques for Endoscopic Ultrasound-Fine Needle Aspiration (EUS-FNA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shyam Varadarajulu (Other)
Responsible Party: Sponsor-Investigator, Shyam Varadarajulu, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F110907002
Record Dates: First submitted 2011-10-18; First posted 2011-12-30 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Pancreatic Tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Biopsy using standard technique of FNA
  Interventions: Procedure: Standard
- Fanning (Other): Biopsy using fanning technique
  Interventions: Procedure: Fanning

INTERVENTIONS:
Procedure: Standard — FNA in a single plane
  Other Names: Standard Versus Fanning Techniques for EUS-FNA
  Arms: Standard
Procedure: Fanning — FNA in multiple planes
  Other Names: Standard Versus Fanning Techniques for EUS-FNA
  Arms: Fanning

SUMMARY:
Endoscopic Ultrasound (EUS)-guided biopsy is the most ideal technique for evaluating a growth in the pancreas. EUS-guided biopsies yield a definitive diagnosis in greater than 80% of cases. In 15-20% of the cases, a definitive diagnosis cannot be made despite multiple attempts. One of the reasons why a diagnosis cannot be made is due to the focal location of the cancer; i.e., the cancer can be situated in a corner of a big mass and the needle fails to sample the cancer cells. The fanning technique is a method where the needle moves in multiple directions within a mass and therefore there is a better chance of the cancer cells being sampled compared to the standard technique where the needle moves in only one direction. The diagnostic performance of both these techniques has not been compared in a randomized fashion.

DETAILED DESCRIPTION:
Fanning technique: Fine Needle Aspiration (FNA) performed in multiple directions within a mass.

Standard technique: FNA performed in unidirectional fashion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years
* Solid Pancreatic Mass Lesions

Exclusion Criteria:

* Age < 19 years
* Coagulopathy
* Unable to consent

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 2 months
  The number of pancreatic masses that are correctly diagnosed with each needle type

SECONDARY OUTCOMES:
Number of passes for diagnosis | 2 months
  Number of passes required to acquire tissue diagnosis using each needle type

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Bang JY, Magee SH, Ramesh J, Trevino JM, Varadarajulu S. Randomized trial comparing fanning with standard technique for endoscopic ultrasound-guided fine-needle aspiration of solid pancreatic mass lesions. Endoscopy. 2013 Jun;45(6):445-50. doi: 10.1055/s-0032-1326268. Epub 2013 Mar 15. PMID 23504490